CLINICAL TRIAL: NCT00408720
Title: Comparison of a Spectral OCT/SLO With the Stratus OCT for Imaging Various Retinal Pathologies
Status: Completed | Type: Observational
Sponsor: The New York Eye & Ear Infirmary (Other)
Other Study IDs: NYEE06-001
Record Dates: First submitted 2006-12-04; First posted 2006-12-07 (Estimated); Last update posted 2006-12-07 (Estimated); Status verified 2006-12

CONDITIONS: Macular Hole; RPE Detachment; Epiretinal Membrane; Posterior Vitreous Detachment
Keywords: Spectral OCT; SLO; Retinal Imagining
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane; Vitreous Detachment

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The purpose of this study is to compare the newly released Spectral OCT/SLO (OTI, Toronto, Canada) with the Zeiss Stratus OCT (Carl-Zeiss Meditec, Dublin, CA) with regards to the quality of the images obtained as well as the ease of use.

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-10; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Rosen, MD, Principal Investigator — New York Eye and Ear Infirmary
Locations (1):
- New York Eye and Ear Infirmary, New York, New York, United States